CLINICAL TRIAL: NCT04010097
Title: Evaluation of Sensitivity, Specificity, Positive and Negative Predictive Values of the Chewing Gum Test for the Diagnosis of Giant Cell Arteritis (Horton's Disease) - ChewingHort
Brief Title: Chewing Gum Test for the Diagnosis of Giant Cell Arteritis (Horton's Disease) - ChewingHort
Acronym: ChewingHort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 87RI19_0009
Record Dates: First submitted 2019-06-27; First posted 2019-07-08 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Horton Disease
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horton group (Experimental): The test involves chewing a chewing gum for 4 minutes plus a standard Horton disease diagnostic
  Interventions: Other: chewing gum
- N Horton Group (Active Comparator): The test involves chewing a chewing gum for 4 minutes
  Interventions: Other: chewing gum

INTERVENTIONS:
Other: chewing gum — The test involves chewing a chewing gum for 4 minutes

SUMMARY:
It is hypothesized that chewing-gums may be a useful test to unmask jaws intermittent claudication in order to enhance the diagnosis of Giant Cell Arteritis (GCA).

DETAILED DESCRIPTION:
GCA is the most common vasculitis. The diagnosis easily could be made in patients over 50 years old with headache, inflammatory belt pain, claudication of the jaws, scalp hyperesthesia, ophthalmological manifestations and an inflammatory syndrome. However, the clinical pictures could be less suggestive, hence diagnostic difficulties. Some patients have only isolated inflammatory syndrome. To confirm the diagnosis, sometimes PET CT or temporal artery biopsy is used, but access to a PET CT is sometimes complex, biopsy of temporal arteries is only positive in about 70% cases. Early diagnosis is important, however, to avoid irreversible complications, especially ophthalmological complications. One in six patients has definitive amaurosis, because of diagnosis delay. The current diagnostic delay is estimated on average at 9 weeks.

Jaw intermittent claudication probably has a very good positive predictive value and this clinical sign often carries conviction. Patients with claudication of the jaws also have a greater visual risk. Kuo reports two observations of patients with claudication of the jaws revealed by the "chewing gum test" after 2 minutes of chewing. It is therefore proposed to perform a chewing gum test to assess the sensitivity and specificity of this test, compared to the interview.

Once the test is done, the study is completed for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Group 1
* Any patient suspected of having GCA, that is to say in practice patients in whom a doctor plans a Doppler ultrasound of temporal arteries or a temporal arteritis biopsy or an imagery (Angio-CT, Angio-MRI, PET- to scan
* Patient over 50 years old
* Patient able to chew a chewing gum for 4 minutes Group 2
* Patients free from GCA
* Age matched (± 3 years)
* Patient able to chew a chewing gum for 4 minutes

Exclusion Criteria:

* Group 1
* Patients known to have a temporomandibular joint pathology
* Patients who started corticosteroid therapy Group 2
* Patients known to have temporomandibular joint pathology
* Patients who started corticosteroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the sensitivity and specificity of the chewing gum test in Horton's disease. | Day 1
  Determination of:
  True positive: Sick people correctly identified as sick False positive: Healthy people incorrectly identified as sick True negative: Healthy people correctly identified as healthy False negative: Sick people incorrectly identified as healthy
  Then wa calculate:
  the number true positives TP the number of false positives FP the number of true negatives TN the number of false negatives.FN
  Specificty= TN/(TN+FP) Sensitivity= : TP/(TP+FN) The test is performed twice an hour apart, to verify its reproducibility, before the introduction of corticosteroid therapy, with chewing gums without sugar.

SECONDARY OUTCOMES:
Evaluate the positive predictive value, the negative predictive value, and the likelihood ratio of the chewing gum test in Horton's disease, | Day1
  predictive value= TP/(TP+FP)

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CH Avignon, Avignon
  - CHU Limoges, Limoges
  - CHU de Nantes, Nantes
  - CH St Antoine, Paris
  - CHU Tours, Tours
  - CH Valenciennes, Valenciennes